CLINICAL TRIAL: NCT05837182
Title: The Role of Augmented Fixation Techniques in Fragility Fracture Pelvis (FFP)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mokhtar Seleem, Principal Investigator, Assiut University
Other Study IDs: augmented fixation in FFP
Record Dates: First submitted 2023-04-06; First posted 2023-05-01 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Fragility Fracture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: augmented fixation techniques — augmented fixation techniques like percutaneous transsarcal screws fixation, tension band plating, INFIX technique, triangular fixation and cement augmentation techniques

SUMMARY:
Assessment of the role of augmented fixation of fragility fracture pelvis in improving functional outcome as a primary outcome and improving union and decreasing mortality and complications as secondary outcomes at 6 months and one year follow up.

DETAILED DESCRIPTION:
During the process of aging, the quality of bones deteriorates making bones more vulnerable for fractures after minor trauma or from normal daily activities. This poor bone quality together with comorbidities increase healing problems and complications and make fixation more difficult. Moreover, immobilization due to fractures has serious complications especially in the elderly. For all theses, fragility fracture-which is defined by WHO as a fracture that is caused by an injury that would be insufficient to fracture normal bones and is the result of reduced compressive and or torsional strength of bone - these fractures have unique criteria making them a special category with its own concerns. One of these fractures is fragility fracture pelvis (FFP) which is expected to triple between 2005 and 2030. This type of fracture has its huge effect on morbidity and mortality of this vulnerable group of people. Due to its special criteria , a new classification system was developed to classify it known as Rommens classification system. This was followed by many literatures focused on this fracture, its morbidity and mortality, role of surgery, minimal invasive techniques and different augmentation fixation techniques, but they did not reach to a clear algorithm for management and did not clearly identify the role of augmented fixation techniques on different outcomes of this fracture . Fixation augmentation techniques which are defined as surgical techniques aimed at increasing implant stability and used in poor bone quality like in geriatric population. the investigators hypothesis is augmented fixation will improve the functional outcomes of fragility fracture pelvis. These techniques may include percutaneous transsarcal screws fixation, tension band plating, INFIX technique, triangular fixation and cement augmentation techniques.

the investigators will try to answer this question which is "what is the effect of augmented fixation techniques on functional outcomes of fragility fracture pelvis? ''.

ELIGIBILITY:
Inclusion Criteria:

1. Patients above age of sixty years.
2. Fragility fracture pelvis
3. injury severity score below 17.
4. Controlled comorbidities

Exclusion Criteria:

1. Malignancy in bony pelvis.
2. Chronic kidney disease on regular dialysis,
3. Skin lesion at admission like Morel-Lavallée lesion.

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: people above age of sixty males and females with fracture pelvis ,not polytraumatized without uncontrolled comorbidities
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-05-06 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
assess change in functional outcome of augmented fixation techniques in fragility fracture pelvis | at 6 weeks, 6 months and one year
  functional outcome using Majeed score system(0 to 100) with 100 is best outcome

SECONDARY OUTCOMES:
assess change in radiological union and complications | X ray at 6 weeks, 6 months and one year one year
  using X ray
assess change in radiological union and complications | CT at 6 months and one year
  using CT
one year mortality rate | one year
  mortality rate at one year

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Seleem, MBBS, Principal Investigator — Assiut University

REFERENCES:
- [Background] Omichi T, Takegami Y, Tokutake K, Saito Y, Ito O, Ando T, Imagama S. Mortality and functional outcomes of fragility fractures of the pelvis by fracture type with conservative treatment: a retrospective, multicenter TRON study. Eur J Trauma Emerg Surg. 2022 Aug;48(4):2897-2904. doi: 10.1007/s00068-021-01839-1. Epub 2021 Dec 1. PMID 34850256
- [Background] Rommens PM, Hofmann A. Fragility fractures of the pelvis. Cham: Springer International Publishing; 2017
- [Background] Rommens PM, Hofmann A. Comprehensive classification of fragility fractures of the pelvic ring: Recommendations for surgical treatment. Injury. 2013 Dec;44(12):1733-44. doi: 10.1016/j.injury.2013.06.023. Epub 2013 Jul 18. PMID 23871193
- [Background] Majeed SA. Grading the outcome of pelvic fractures. J Bone Joint Surg Br. 1989 Mar;71(2):304-6. doi: 10.1302/0301-620X.71B2.2925751.
- [Background] Kulakowski M, Reichert P, Elster K, Sleczka P, Oleksy L, Krolikowska A. Safety and efficacy of two ilioiliac tension band plates osteosynthesis of fragility fractures of the pelvis. Sci Rep. 2022 Nov 28;12(1):20436. doi: 10.1038/s41598-022-24525-7. PMID 36443346
- [Background] Haveman RA, Baumlein M, van Veelen N, Oberkircher L, Beeres FJP, Babst R, Ruchholtz S, Link BC. Percutaneous sacroiliac screw fixation in fragility fractures of the pelvis: Comparison of two different augmentation techniques. Injury. 2022 Dec;53(12):4062-4066. doi: 10.1016/j.injury.2022.09.050. Epub 2022 Oct 8. PMID 36220693
- [Background] Rommens PM, Hofmann A, Kraemer S, Kisilak M, Boudissa M, Wagner D. Operative treatment of fragility fractures of the pelvis: a critical analysis of 140 patients. Eur J Trauma Emerg Surg. 2022 Aug;48(4):2881-2896. doi: 10.1007/s00068-021-01799-6. Epub 2021 Oct 11. PMID 34635938